CLINICAL TRIAL: NCT04593680
Title: Institute of HIV Research and Innovation (IHRI)
Brief Title: Assessment of Drug-drug Interactions Between Masculinizing Hormone Therapy and Antiretroviral Agents Concomitantly for Pre-exposure Prophylaxis Among Transgender Men
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thai Red Cross AIDS Research Centre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: iMACT
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Emtricitabine; Tenofovir; tenofovir alafenamide

STUDY DESIGN:
Masking Description: An open-label, randomized, two-arm prospective PK study of HIV-negative TGM taking MHT and daily PrEP:
  Arm 1: Twenty HIV-negative TGM will take daily TDF/FTC-based PrEP
  Arm 2: Twenty HIV-negative TGM will take daily F/TAF-based PrEP
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20 HIV-negative TGM will take daily TDF/FTC-based PrEP (Experimental): MHT will be initiated on week 0 and will be last administered on week 12. PrEP will be initiated on week 6 and continued without interruption.
  MHT: Intramuscular testosterone enanthate 200 mg bi-weekly, which is the treatment of choice for MHT in the Pribta Clinic, will be provided to all participants.
  PrEP: Fixed-dose combination of emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg (F/TDF) and emtricitabine 200 mg/tenofovir alafenamide 25 mg (F/TAF) will be provided for arm 1 and 2, respectively.
  Pharmacokinetic measurement of study drug Two full pharmacokinetic (PK) measurements will be performed. Samples collected will include: plasma for testosterone, emtricitabine (FTC) and tenofovir (TFV), with an additional tenofovir alafenamide (TAF).
  Interventions: Drug: Emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg (F/TDF) and emtricitabine 200 mg/tenofovir alafenamide 25 mg (F/TAF)
- 20 HIV-negative TGM will take daily F/TAF-based PrEP (Experimental): MHT will be initiated on week 0 and will be last administered on week 12. PrEP will be initiated on week 6 and continued without interruption.
  MHT: Intramuscular testosterone enanthate 200 mg bi-weekly, which is the treatment of choice for MHT in the Pribta Clinic, will be provided to all participants.
  PrEP: Fixed-dose combination of emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg (F/TDF) and emtricitabine 200 mg/tenofovir alafenamide 25 mg (F/TAF) will be provided for arm 1 and 2, respectively.
  Pharmacokinetic measurement of study drug Two full pharmacokinetic (PK) measurements will be performed. Samples collected will include: arm 2, measurement; and peripheral blood mononuclear cells (PBMC) for emtricitabine-triphosphate (FTC-TP) and tenofovir-diphosphate (TFV-DP) intracellular quantification.
  Interventions: Drug: Emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg (F/TDF) and emtricitabine 200 mg/tenofovir alafenamide 25 mg (F/TAF)

INTERVENTIONS:
Drug: Emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg (F/TDF) and emtricitabine 200 mg/tenofovir alafenamide 25 mg (F/TAF) — The first full PK measurement of MHT will be performed starting at week 4 and end at week 6 to assess the steady-state plasma PK of testosterone in the absence of PrEP. The second PK measurement of MHT will be performed starting at week 12 and end at week 14 to assess plasma PK of testosterone in the presence of both MHT and PrEP. The first full PK measurement of PrEP will be performed at week 12 to assess the steady-state plasma PK of FTC, TFV, and TAF; and intracellular PBMC FTC-TP and TFV-DP in the presence of both MHT and PrEP. The second measurement of PrEP will be performed at week 16 to assess plasma PK of FTC, TFV, and TAF; and intracellular PBMC FTC-TP and TFV-DP in the absence of MHT.

SUMMARY:
There are currently no published studies addressing drug-drug interactions (DDI) between masculinizing hormone therapy (MHT) and pre-exposure prophylaxis (PrEP) among transgender men (TGM). This could lead to concerns and subsequent prioritizing MHT over PrEP among TGM. Because tenofovir alafenamide (TAF) can achieve higher intracellular tenofovir diphosphate (TFV-DP) levels with lower tenofovir plasma concentrations, it is promising that both plasma tenofovir (TFV) and intracellular TFV-DP levels might not be significantly affected by MHT. The current study aims to determine the pharmacokinetics (PK) DDI between MHT and daily PrEP among TGM.

ELIGIBILITY:
Inclusion Criteria:

1. Thai nationality
2. Age 18-40 years old
3. Female-to-Male transgender individual
4. HIV-negative
5. Body mass index 18.5-24.9 kg/m2
6. Negative urine pregnancy test
7. Calculated creatinine clearance (CrCl) ≥60 mL/min, as estimated by the Cockcroft-Gault equation
8. Alanine aminotransferase (ALT) ≤2.5 x ULN
9. Signed the informed consent form

Exclusion Criteria:

1. Known history of allergy to hormonal component to be used in the study
2. Use of pre-exposure prophylaxis or post-exposure prophylaxis in the past 30 days
3. Use of injectable MHT in the past 3 months
4. Evidence of current hepatitis B virus infection (HBV) - i.e. hepatitis B surface antigen [HBsAg] positive
5. Evidence of current hepatitis C virus infection (HCV) - i.e. HCV antibody positive
6. History of myocardial infarction or coronary artery disease
7. Current use of any of the following:

   * Anticonvulsants: carbamazepine, oxcarbazepine, phenytoin, or phenobarbital
   * Herbs: gingko biloba, St John's wort or milk thistle
   * Anti-infective agents: protease inhibitors, rifampicin or rifabutin
8. History of gastrointestinal tract surgery that alter gastrointestinal tract and/or drug absorption
9. Alcohol or drug use that, in the opinion of the investigator, would interfere with completion of study procedures

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma TFV level | 2 years
  1. Changes in plasma testosterone levels [Time Frame: Measured at week 4 and week 12 of the study period]
  2. Changes in plasma TFV levels [Time Frame: Measured at week 12 and week 16 of the study period]
  3. Changes in plasma emtricitabine (FTC) levels [Time Frame: Measured at week 12 and week 16 of the study period]
  4. Changes in plasma TAF levels [Time Frame: Measured at week 12 and week 16 of the study period]
  5. Changes in peripheral blood mononuclear cell TFV-DP levels [Time Frame: Measured at week 12 and week 16 of the study period]
  6. Changes in peripheral blood mononuclear cell (PBMC) emtricitabine triphosphate (FTC-TP) levels [Time Frame: Measured at week 12 and week 16 of the study period]

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of HIV Research and Innovation (IHRI), Bangkok, Pathumwan, Thailand

REFERENCES:
- [Derived] Hiransuthikul A, Thammajaruk N, Kerr S, Janamnuaysook R, Nonenoy S, Hongchookiat P, Trichavaroj R, Tawon Y, Boonruang J, Teeratakulpisarn N, Cressey TR, Anderson PL, Phanuphak N; iMACT study team. Exploring potential drug-drug interactions between masculinizing hormone therapy and oral pre-exposure prophylaxis (F/TDF and F/TAF) among transgender men (iMACT study): a randomized, open-label pharmacokinetic study in Thailand. J Int AIDS Soc. 2025 Apr;28(4):e26445. doi: 10.1002/jia2.26445. PMID 40195242